CLINICAL TRIAL: NCT04949386
Title: A Randomized, Placebo-Controlled Phase II Study To Evaluate The Safety, Tolerability And Efficacy Of S-1226 In Post-Covid-19 Subjects With Persistent Respiratory Symptoms.
Brief Title: Safety, Tolerability and Efficacy of S-1226 in Post-COVID-19 Subjects With Persistent Respiratory Symptoms.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SolAeroMed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAMi-06-1-01
Record Dates: First submitted 2021-06-30; First posted 2021-07-02 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Post Acute COVID-19 Syndrome; Long COVID; COVID-19 Respiratory Infection
Keywords: S-1226; Prolonged post viral respiratory symptoms
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — perfluorooctylbromide and CO2 drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with S-1226 (8%) (Experimental): Subjects randomized to this treatment arm will receive S-1226(8%) twice daily for 7 consecutive days. S-1226 will be administered by inhalation for 3-4 minutes.
  Interventions: Drug: S-1226 (8%)
- Placebo (Placebo Comparator): Subjects randomized to receive placebo will be administered with medical grade air with 3ml saline (0.9% NaCl) using the Circulaire II hybrid system. Placebo will be administered by inhalation for 3-4 minutes.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: S-1226 (8%) — S-1226 has two components delivered by inhalation. It is a mixture of perfluorooctylbromide (PFOB) delivered in gas/aerosol/vapor form within a medical gas mixture containing 8% CO2.
  Other Names: S-1226
  Arms: Treatment with S-1226 (8%)
Other: Placebo — Placebo will delivered by inhalation of saline (0.9% NaCl) and Medical grade air.
  Arms: Placebo

SUMMARY:
This is a randomized (1:1) , placebo-controlled phase II study to evaluate the safety, tolerability and efficacy of S-1226 in Post-COVID-19 subjects (n≤48) with persistent respiratory symptoms. Subjects will receive twice daily treatments of either Placebo or S-1226 (8%) for 7 days.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, phase II proof of concept study to evaluate the safety, tolerability and efficacy of S-1226 in Post-COVID-19 subjects (n≤48) with persistent respiratory symptoms.

S-1226 contains a potent, safe and well-tolerated bronchodilator gas (extrinsic carbon dioxide or CO2) and perflubron (PFOB), a synthetic surfactant that facilitates restoration of surfactant function and mucus clearance. The inhaled S-1226 combination of gas, vapor and liquid aerosol penetrates obstructed airways, resulting in rapid bronchodilation, enhanced blood oxygenation, improved mucus clearance and reduction of work of breathing.

Primary objective of this study is to evaluate the safety and tolerability of S-1226 composed of perflubron with 8% carbon dioxide in subjects with persistent post acute COVID-19 respiratory symptoms. The secondary objective is to establish proof of concept that S-1226 is effective in normalizing lung symptoms, including cough, breathlessness and lung function in subjects with persistent post-acute COVID-19 respiratory symptoms.

The study will consist of three parts: screening and randomization period, Treatment and evaluation, follow up period.

1. Screening, and randomization: subjects will be randomized (1:1) to either receive placebo or S-1226 treatment.
2. Treatment and evaluation period: subjects will receive either placebo -medical grade air with 3ml saline (0.9% NaCl) - or S-1226 (8% CO2) for 7 days twice daily. A single dose of S1226 (8%) will be administered over 3-4 minutes at each visit. Subjects will have the option to receive at home treatments once they been trained and verified as competent in handling study equipment.
3. A follow up period 7 days after final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the following criteria to be included in the study:

  1. Male or Females between 18 -80 years of age at the time of consent
  2. Able to provide informed consent.
  3. Prior confirmed COVID-19 diagnosis by standard Real time Polymerase Chain Reaction (RT-PCR) assay or Immunoglobin M/G (IgM/IgG) rapid serological test at least 4 weeks prior to screening visit.
  4. Ambulatory patients may be attending COVID long term follow up clinic or discharged from hospital for at least one week.
  5. Evidence of new and/or persistent respiratory symptoms at least 4 weeks after the onset of acute COVID-19 infection. This will be determined by history of respiratory symptoms: cough, wheeze, limitation of activities.
  6. Able to perform an exercise of moderate activity e.g., walking up a hill or climbing stairs (required to assess Borg RPE)
  7. Able to walk unaided for a minimum distance of 10 meters (distance validated for completion of 6-minute walk test)

Exclusion Criteria:

* Subjects to whom any of the following applies will be excluded from the study:

  1. Pregnancy or of childbearing age without a highly effective method or at least two forms of effective contraception and/ or abstinence for the duration of study. Highly effective methods of contraception (Contraception with < 1% failure rate) are: hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation. Effective methods of contraception may include barrier methods of contraception (e.g., male condom, female condom, cervical cap, diaphragm, contraceptive sponge).
  2. Breastfeeding females.
  3. Evidence of active thromboembolic disorder - defined by those receiving parenteral anticoagulant or thrombolytic therapy.
  4. Pre-existing evidence of unstable angina and myocardial infraction during the previous month, contraindications to the 6MWT.
  5. Subject, who in the opinion of the Investigator, is unsuitable to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Effects | 16 days
  The number and percent of treatment emergent adverse events will be monitored, recorded and graded for severity and assigned attribution. The severity will be assessed in the following manner:
  Mild: Awareness of signs or symptoms, but are easily tolerated and are of minor irritant type, causing no limitations of usual activities. Signs or symptoms may require minor action or additional therapy.
  Moderate: Discomfort severe enough to cause some limitations of usual activities and may require action or additional therapy.
  Severe: Incapacitating with inability to carry out usual activities and requires specific action and/or medical attention. Note: the term severe is not the same as "serious", which is based on subject/event outcome or action criteria usually associated with events that pose a threat to a subject's life or functioning. Seriousness (not severity) serves as a guide for defining regulatory reporting obligations.

SECONDARY OUTCOMES:
Normalization in 6-minute walk test (6MWT) distance | 16 days
  Changes in induced shortness of breath will be monitored using the 6 Minute walk test (6MWT) with continuous oxygen saturation (SpO2) monitoring . Normalization will be assessed by a return to normal distance values established in the literature.
Changes in percent predicted forced expiratory volume in 1 second | 16 days
  Change from baseline in percent of predicted forced expiratory volume in 1 Second (FEV1) will be calculated by measuring FEV1 at baseline and after treatment. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Changes in from baseline in respiratory symptoms assessed by the St George's Respiratory Questionnaire (SGRQ). | 16 days
  St George's Respiratory Questionnaire (SGRQ), a two-part questionnaire that evaluates participant symptoms, including cough, (part 1) and activities and impact (part 2). Scores range from 0 to100 with higher scores indicating more limitations/perceived distress. Scores will be compared to the established minimally clinically important difference (MCID).

OTHER OUTCOMES:
Change from baseline in Forced Vital Capacity. | 16 days
  Change from baseline in Forced Vital Capacity (FVC) will be measured. FVC is the total volume of air that can be exhaled during a maximal forced expiration effort.
Changes from baseline in Diffusing Lung Capacity | 16 days
  Changes from Baseline in Diffusing lung capacity (DLCO) will be measures. DLCO is a measurement used to evaluate the lungs ability to transfer gas from inspired air to the bloodstream.
Changes from baseline in Oxygen Saturation (SpO2) | 16 days
  Changes from baseline in percent of oxygen saturation (measured by pulse oximetry) will be calculated by measuring oxygen saturation before and up to 30 minutes after treatment.
Changes in from baseline in respiratory symptoms assessed by the modified Medical Research Council (mMRC) scale of dyspnea during daily activity. | 16 days
  The modified Medical Research Council (mMRC) scale of dyspnea used assess baseline and subsequent activity related dyspnea. Scores range from 0-4, with increasing scores representing greater difficulty in performing daily activities.
Changes in from baseline in respiratory symptoms assessed by the Borg Rating of Perceived Exertion (RPE) for dyspnea during exertion. | 16 days
  Borg Rating of Perceived Exertion (RPE) a categorical scale used to assess dyspnea during exertion. The lowest score, 6, represents No exertion/effort at all while the highest score of 20 represents absolute maximal effort/exhaustion.
Changes in from baseline in respiratory symptoms assessed by Visual Analogue Scale (VAS) for dyspnea while at rest. | 16 days
  A 10 cm Visual Analogue Scale (VAS) to assess participant dyspnea while at rest at the time of Assessment. Three delineations will be placed on the scale (0 being no dyspnea, 5 (middle) and 10 being max dyspnea) for participants to mark with a cross.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Montgomery, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swystun V, Green FHY, Dennis JH, Rampakakis E, Lalli G, Fadayomi M, Chiu A, Shrestha G, El Shahat SG, Nelson DE, El Mays TY, Pieron CA, Leigh R. A phase IIa proof-of-concept, placebo-controlled, randomized, double-blind, crossover, single-dose clinical trial of a new class of bronchodilator for acute asthma. Trials. 2018 Jun 18;19(1):321. doi: 10.1186/s13063-018-2720-6. PMID 29914544
- [Background] Green FH, Leigh R, Fadayomi M, Lalli G, Chiu A, Shrestha G, ElShahat SG, Nelson DE, El Mays TY, Pieron CA, Dennis JH. A phase I, placebo-controlled, randomized, double-blind, single ascending dose-ranging study to evaluate the safety and tolerability of a novel biophysical bronchodilator (S-1226) administered by nebulization in healthy volunteers. Trials. 2016 Jul 28;17:361. doi: 10.1186/s13063-016-1489-8. PMID 27464582
- [Background] El Mays TY, Choudhury P, Leigh R, Koumoundouros E, Van der Velden J, Shrestha G, Pieron CA, Dennis JH, Green FH, Snibson KJ. Nebulized perflubron and carbon dioxide rapidly dilate constricted airways in an ovine model of allergic asthma. Respir Res. 2014 Sep 16;15(1):98. doi: 10.1186/s12931-014-0098-x. PMID 25355286